CLINICAL TRIAL: NCT00703209
Title: Controlled, Randomized, Double-Blinded, Prospective Study On the Role of Decompression of Lower Extremity Nerves for the Treatment of Patients With Symptomatic Diabetic Neuropathy With Chronic Nerve Compression
Brief Title: Study on the Role of Decompression of Lower Extremity Nerves for the Treatment of Patients With Symptomatic Diabetic Neuropathy With Chronic Nerve Compression
Acronym: DNND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Shai Michael Rozen, Associate Professor, Department of Plastic Surgery, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UTSW-001
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Painful Diabetic Neuropathy
Keywords: symptomatic diabetic neuropathy; diabetes; burning feet; Diabetic Neuropathy; Loss of sensation in the foot; Neuropathy; Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients who are randomized to receive surgical care, will receive the nerve decompression, along with similar incisions on the opposite leg, but no decompression on that leg. This will serve as the patient's control leg, and also blind them to the treatment leg.
  Interventions: Procedure: Nerve Decompression
- 2 (No Intervention): Subjects who are not randomized to receive the surgical procedure will be followed up with the same clinic visits as the patients who are receiving the surgical procedure.

INTERVENTIONS:
Procedure: Nerve Decompression — Nerve decompression on a randomized leg, with similar skin incisions on the opposite leg so that the patient is "blinded" to which leg received the decompression.
  Arms: 1

SUMMARY:
The UT Southwestern Medical Center at Dallas would like to give you information about a research study that is being done for patients with painful diabetic neuropathy and have not responded to medical treatment. Doctors from the departments of Internal Medicine, Physical Medicine and Rehabilitation, Neurology, Pain Management and Plastic Surgery are conducting a research study to examine the effects of nerve decompression on decreasing the pain associated with diabetic neuropathy and increasing the sensation at the bottom of the foot.

DETAILED DESCRIPTION:
Dr. Shai Rozen, is working with physicians from Internal Medicine, Neurology, and Physical Medicine and Rehabilitation to conduct a clinical study on patients with painful diabetic neuropathy. Specifically, regarding the efficacy of peripheral nerve decompression in the lower extremity in a select group of patients which may have superimposed nerve compression in addition to their diabetic neuropathy. Initial data supports success rates at around 80% in terms of significant alleviation of pain and restoration of at least protective sensation and long term follow ups have suggested decrease in prevalence of infections, ulcerations, and amputations.

Potential candidates for the study are patients who have symptomatic painful diabetic neuropathy who have not responded to medical treatment (glucose control, pain medications)and continue to have severe pain.

It is thought today that one third of patients with diabetic neuropathy may have superimposed nerve compression in the nerves in the leg, or in other words the nerves may be pressed by the surrounding tissue. This nerve compression is what might be contributing to the pain, and often loss of sensation at the bottom of your feet. The principle is similar to carpal tunnel syndrome which is pressure of a nerve in the wrist. Carpal tunnel syndrome is seen in 14-30% of patients with diabetes compared to 2% in the general population.

This study involves one year of close care and follow-up. As a part of this study, you will have regular evaluations by a foot care specialist from Physical Medicine and Rehabilitation, receive glucose management tips from a Diabetic Nurse Educator, and also have specialized, non-invasive testing in the Neurology department. The care that you would receive for being a part of this study is highly exceptional due to the various departments involved and their dedication to this research.

Initial data supports success rates at around 80% in terms of significant alleviation of pain and restoration of at least protective sensation and long term follow ups have suggested decrease in prevalence of infections, ulcerations, and amputations.

Potential candidates for the study are patients who have symptomatic painful diabetic neuropathy who have not responded to medical treatment (glucose control, pain medications) for at least one year and continue to have severe pain.

Dr. Shai Rozen is the principal investigator on this study, and Julia Kalayanamit is the clinical coordinator. We are both very happy to speak with you if you would like more information about the study, including appointments, scheduling and visit activities.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 Diabetes
* Diagnosed with peripheral neuropathy
* Symptoms of: pain and/or numbness
* Bilateral symptoms (pain in both legs)
* Have been treated non-surgically
* Aged 18-80
* All genders and all races

Exclusion Criteria:

* Cardiac or renal pedal edema
* Medical condition which does not allow surgery
* Inadequate glycemic control
* Skin ulcer
* Charcot's foot
* Symptoms of radiculopathy/sciatic-type nerve pain
* Inadequate nutrient circulation in the feet
* Weight greater than 300 lbs.
* Psychiatric problems or alcohol/drug abuse
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2008-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To determine if nerve decompression of lower extremities in patients suffering from painful symptomatic diabetic neuropathy with chronic nerve compression, has a significant impact on alleviation of pain, and improvement in quality of life. | 2 years

SECONDARY OUTCOMES:
To measure changes in quality of life. This includes medication changes, pain relief, restoration of sensation, etc. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shai M Rozen, MD, Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States